CLINICAL TRIAL: NCT05422976
Title: Safety and Tolerability of a Single Intra-articular Highly Concentrated Hyaluronic Acid Injection in the Treatment of Symptomatic Knee Osteoarthritis : Pilot, 6-months, Open-label, Single-arm Investigation
Brief Title: EVI-01-IT Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aptissen SA (Industry)
Collaborators: Donawa Lifescience (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVI-01-IT
Record Dates: First submitted 2022-06-07; First posted 2022-06-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: highly concentrated hyaluronic acid; knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EVI-01 treatment (Experimental): EVI-01 should be injected within the synovial cavity using standard procedures for intra-articular (IA) injections by a physician skilled in performing IA injections.
  Interventions: Device: EVI-01

INTERVENTIONS:
Device: EVI-01 — High molecular weight Hyaluronic Acid

SUMMARY:
Prospective, single arm, pilot study to assess the safety and tolerability of a single intra-articular injection of EVI-01 for the treatment of symptomatic knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen (18) years old or above;
* Patient signed informed consent form;
* Patients with stable symptoms related to knee osteoarthritis for at least 3 months prior to screening;
* Failure, inadequate response or intolerance to analgesics and/or NSAIDs or low-grade opioids;
* Kellgren-Lawrence radiographic stage: II-III diagnosed in the previous 12 months;
* WOMAC average pain index score > 40 mm and < 90 (on a VAS 0-100 mm) on the knee to be treated;
* Difference ≥ 10 mm between the WOMAC average pain score of the knee to be treated and WOMAC average pain score of the contralateral knee at screening;
* Body Mass Index (BMI) inferior to 35 kg/m2 (weight/height).

Exclusion Criteria:

* Concomitant inflammatory joint disorder;
* Had received previous visco-supplementation treatment in the study knee within 6 months or intra articular corticosteroids within 3 months* prior to inclusion;
* Infection in or around the study knee;
* Relevant skin disease in the area of injection site;
* Documented presence of injury or trauma of the study knee at screening, including evidence of a subchondral fracture, meniscal lesion, presence of bone or cartilage fragments in the study knee;
* History of allergy or intolerance to sodium hyaluronate;
* Documented presence of osteonecrosis in one or both knees;
* Inability to understand the study procedure;
* Participation in another clinical trial within 30 days prior to screening;
* Ongoing therapy with daily dosage > 101 mg of acetylsalicylic acid as part of cardiovascular preventive treatment. If dose < 101 mg, it must be maintained during the study;
* Pregnant or breast-feeding at inclusion.

  * 1 month = 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 6 months
  Primary objective of this study is to assess the safety and tolerability of EVI-01 following single intraarticular administration in the knee joint, assessed with adverse events monitoring throughout the follow up duration of six months.

SECONDARY OUTCOMES:
Change in patient-reported pain intensity | 7 days
  Change in patient-reported pain intensity at Days 1 to 7 compared to baseline will be assess using a 0-100 mm Visual Analogue Scale (VAS), in which 0 means ''no pain at all'' and 100 means ''the worst possible pain''.
Change in WOMAC index | 6 months
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) consists of a total of 24 questions divided in 5 questions related to pain, 2 questions related to stiffness and 17 questions related to difficulties in performing activities of daily living in relation to physical function. Each question refers to a 0-100 mm Visual Analogue Scale (VAS) in which 0 means ''no pain at all'' and 100 means ''the worst possible pain''. Change in WOMAC pain, stiffness, function and total score will be assess using WOMAC index at Day 7, Day 14, Day 30, Day 90 and Day 180 compared to baseline
Patient satisfaction for the overall treatment effect | 6 months
  Measurements of relief satisfaction by the patient will be assess using a 7 points Likert scale at Day 180. A 7 point Likert scale offers 7 different answer options related to an agreement that would be distinct enough for the respondents (Very good, Good, Fairly good, Same as before, Fairly bad, Bad, Very bad).
Physician satisfaction for the overall treatment effect | 6 months
  Measurements of relief satisfaction by the physician will be assess using a 7 points Likert scale at Day 180. A 7 point Likert scale offers 7 different answer options related to an agreement that would be distinct enough for the respondents (Very good, Good, Fairly good, Same as before, Fairly bad, Bad, Very bad).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, MD, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy